CLINICAL TRIAL: NCT07203690
Title: Development and Application of AI-Based Therapeutic Strategies for Esophageal Cancer Integrating Multimodal Imaging and Digital Pathology
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Xinyang Central Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Qujinrong, Clinical Professor, Henan Cancer Hospital
Other Study IDs: 2025-066
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multimodal AI Esophageal Carcinoma Cohort Protocol: Efficacy and Prognosis of Different Treatment Modalities for Esophageal Squamous Cell Carcinoma

SUMMARY:
The purpose of this clinical study is to conduct a multi-center, big data study to create a neural network decision model for predicting treatment efficacy and prognosis based on multi-modal, multi-temporal imaging features combined with tumor microenvironment scores. It will also use various model interpretation techniques to clarify the role and mechanism of key biomarkers or strongly associated biomarker groups in treatment efficacy and prognosis. Ultimately, it aims to achieve the research and application of AI treatment strategies combining multi-modal imaging and digital pathology to guide clinicians in the personalized treatment strategies for patients with esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Histologically confirmed esophageal carcinoma by biopsy;
3. No prior antitumor therapy received.

Exclusion Criteria:

1. Contraindications to MRI examination;
2. Poor compliance with antitumor therapy;
3. Unwillingness to participate in the study;
4. Image quality inadequate for diagnostic requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll 7,000 esophageal carcinoma patients from multiple centers. Participants will receive CT and mpMRI scans before, during, and after treatment, as required for evaluating surgery, neoadjuvant therapy, or definitive chemoradiation. PET-CT will be performed if distant metastasis is suspected. Whole-slide digital scanning will be applied to biopsy and surgical specimens for pathological analysis.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | January 2025 - December 2027
  The proportion of patients achieving pathological complete response (ypT0 ypN0) after neoadjuvant therapy.
Overall Survival (OS) | January 2025 - December 2027
  The time from treatment initiation to death from any cause.
Event-Free Survival (EFS) | January 2025 - December 2027
  The time from treatment initiation to disease progression, recurrence, new primary cancer, or death.
Disease-Free Survival (DFS) | January 2025 - December 2027
  The time from curative-intent surgery to disease recurrence or death.

IPD SHARING:
Plan to Share IPD: Undecided